CLINICAL TRIAL: NCT01845740
Title: A Phase Ib Study of Milatuzumab Administered Subcutaneously in Patients With Active Systemic Lupus Erythematosus (SLE)
Brief Title: Phase Ib Study of SC Milatuzumab in SLE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMMU-115-04
Record Dates: First submitted 2013-04-17; First posted 2013-05-03 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-02

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic; Lupus Vasculitis, Central Nervous System; Lupus Nephritis
Keywords: systemic lupus erythematoses; lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic; Lupus Vasculitis, Central Nervous System; Lupus Nephritis | interventions — milatuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milatuzumab SC 250 mg (Experimental): Milatuzumab 250 mg will be administered subcutaneously once weekly for 4 weeks.
  Interventions: Drug: milatuzumab
- Milatuzumab 150 mg SC (Experimental): Milatuzumab 150 mg will be administered subcutaneously once weekly for 4 weeks.
  Interventions: Drug: milatuzumab
- Placebo SC (Placebo Comparator): Placebo will be administered subcutaneously once weekly for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: milatuzumab — Milatuzumab has been used in clinical trials for multiple myeloma, non-Hodgkin's lymphoma and leukemia in the intravenous dosing form. In this study, milatuzumab is being given subcutaneously in patients with lupus.
  Other Names: Milatuzumab is a Cd74 targeted humanized monoclonal antibody.
  Arms: Milatuzumab 150 mg SC; Milatuzumab SC 250 mg
Drug: Placebo — Placebo will be administered subcutaneously once weekly for 4 weeks.
  Arms: Placebo SC

SUMMARY:
Milatuzumab will be given subcutaneously at different dose levels once (depending on the dose level) for 4 weeks to determine if milatuzumab helps to control lupus (SLE).

DETAILED DESCRIPTION:
Milatuzumab or placebo will be given subcutaneously once weekly for 4 weeks to determine if milatuzumab helps to control lupus (SLE). The treatment portion of the study lasts 4 weeks. Then patients are followed for disease activity for at least 12 weeks. If patients respond to the study drug, they may be eligible for one course of retreatment, again followed by 12 weeks of follow-up. Patients who showed a response will continue to be followed at timepoints up to one year after treatment to assess how long the response lasts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years old
* Signed written informed consent before study entry
* Diagnosis of SLE by American College of Rheumatology revised criteria (meets ≥ 4 criteria)
* Positive ANA (titer ≥ 1:80) at study entry
* At least 1 BILAG A or 2 BILAG B scores in any organ/body system and ≥ 6 SELENA-SLEDAI score
* Receiving at least 5.0 mg/day oral prednisone (or equivalent) at stable doses for at least 4 weeks prior to study entry
* If receiving immunosuppressives or antimalarial agents, at stable doses for at least 4 weeks prior to study entry

Exclusion Criteria:

* Pregnant or lactating women. Women of childbearing potential must have a negative pregnancy test.
* Women of childbearing potential and fertile men not practicing or unwilling to practice birth control during the study
* Rituximab, belimumab, other prior antibody, investigational or experimental therapy within 6 months
* Allergic to murine, chimeric, humanized or human antibodies
* Hematologic abnormalities not attributed to lupus: hemoglobin < 8.0 mg/dL, WBC < 2000/L, ANC < 1500/L, platelets < 50,000/L,
* AST, ALT or alkaline phosphatase > 3 times upper limit of normal and not attributed to lupus
* Serum creatinine > 2.5 mg/dL, proteinuria > 3.5 g/day
* Received live vaccine within 4 weeks
* Thrombosis, spontaneous or induced abortion, stillbirth or live birth within 4 weeks
* Antiphospholipid antibodies AND a history of thromboembolic events
* On oral anticoagulants (not including NSAIDs) within 4 weeks
* Active infection with antibiotics within 7 days
* Infection requiring hospitalization or herpes zoster treatment within 4 weeks
* Long-term infectious diseases (tuberculosis, fungal infections) active within 2 years
* Malignancy (except squamous or basal cell carcinoma, cervical CIS) within 3 years (unless approved by the medical monitor)
* History of recurrent abortions (2 or more)
* Known HIV, hepatitis B or C, other immunosuppressive states
* Other concurrent medical conditions that, in the investigator's opinion, could affect the patient's ability to tolerate or complete the study will not be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | up to 2 years
  Will be assessed using laboratory and clinical data comparing baseline lab results and clinical condition to the lab results and clinical condition/adverse events during treatment and follow-up timepoints up to 2 years.
Obtain preliminary evidence of efficacy for patients with active disease. | up to 2 years
  Will be assessed using the BILAG scoring model for lupus disease activity and symptoms by comparing baseline BILAG measurements against the BILAG measurements obtained during treatment and during follow-up for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, PhD, MD, Principal Investigator — Gilead Sciences
Locations (1):
- Cedars Sinai Medical Center-Wallace Rheumatic Study Center, West Hollywood, California, United States

REFERENCES:
- [Background] Frolich D, Blassfeld D, Reiter K, Giesecke C, Daridon C, Mei HE, Burmester GR, Goldenberg DM, Salama A, Dorner T. The anti-CD74 humanized monoclonal antibody, milatuzumab, which targets the invariant chain of MHC II complexes, alters B-cell proliferation, migration, and adhesion molecule expression. Arthritis Res Ther. 2012 Mar 9;14(2):R54. doi: 10.1186/ar3767. PMID 22404985
- [Background] Gupta P, Goldenberg DM, Rossi EA, Cardillo TM, Byrd JC, Muthusamy N, Furman RR, Chang CH. Dual-targeting immunotherapy of lymphoma: potent cytotoxicity of anti-CD20/CD74 bispecific antibodies in mantle cell and other lymphomas. Blood. 2012 Apr 19;119(16):3767-78. doi: 10.1182/blood-2011-09-381988. Epub 2012 Jan 23. PMID 22271448
- [Background] Alinari L, Mahoney E, Patton J, Zhang X, Huynh L, Earl CT, Mani R, Mao Y, Yu B, Quinion C, Towns WH, Chen CS, Goldenberg DM, Blum KA, Byrd JC, Muthusamy N, Praetorius-Ibba M, Baiocchi RA. FTY720 increases CD74 expression and sensitizes mantle cell lymphoma cells to milatuzumab-mediated cell death. Blood. 2011 Dec 22;118(26):6893-903. doi: 10.1182/blood-2011-06-363879. Epub 2011 Oct 31. PMID 22042694
- [Background] Santana JM, Grellier P, Rodier MH, Schrevel J, Teixeira A. Purification and characterization of a new 120 kDa alkaline proteinase of Trypanosoma cruzi. Biochem Biophys Res Commun. 1992 Sep 30;187(3):1466-73. doi: 10.1016/0006-291x(92)90467-y. PMID 1417823
- [Background] Alinari L, Yu B, Christian BA, Yan F, Shin J, Lapalombella R, Hertlein E, Lustberg ME, Quinion C, Zhang X, Lozanski G, Muthusamy N, Praetorius-Ibba M, O'Connor OA, Goldenberg DM, Byrd JC, Blum KA, Baiocchi RA. Combination anti-CD74 (milatuzumab) and anti-CD20 (rituximab) monoclonal antibody therapy has in vitro and in vivo activity in mantle cell lymphoma. Blood. 2011 Apr 28;117(17):4530-41. doi: 10.1182/blood-2010-08-303354. Epub 2011 Jan 12. PMID 21228331
- [Background] Hertlein E, Triantafillou G, Sass EJ, Hessler JD, Zhang X, Jarjoura D, Lucas DM, Muthusamy N, Goldenberg DM, Lee RJ, Byrd JC. Milatuzumab immunoliposomes induce cell death in CLL by promoting accumulation of CD74 on the surface of B cells. Blood. 2010 Oct 7;116(14):2554-8. doi: 10.1182/blood-2009-11-253203. Epub 2010 Jun 23. PMID 20574049
- [Background] Berkova Z, Tao RH, Samaniego F. Milatuzumab - a promising new immunotherapeutic agent. Expert Opin Investig Drugs. 2010 Jan;19(1):141-9. doi: 10.1517/13543780903463854. PMID 19968579
- [Background] Stein R, Smith MR, Chen S, Zalath M, Goldenberg DM. Combining milatuzumab with bortezomib, doxorubicin, or dexamethasone improves responses in multiple myeloma cell lines. Clin Cancer Res. 2009 Apr 15;15(8):2808-17. doi: 10.1158/1078-0432.CCR-08-1953. Epub 2009 Apr 7. PMID 19351768
- [Background] Mark T, Martin P, Leonard JP, Niesvizky R. Milatuzumab: a promising new agent for the treatment of lymphoid malignancies. Expert Opin Investig Drugs. 2009 Jan;18(1):99-104. doi: 10.1517/13543780802636162. PMID 19053886
- [Background] Stein R, Mattes MJ, Cardillo TM, Hansen HJ, Chang CH, Burton J, Govindan S, Goldenberg DM. CD74: a new candidate target for the immunotherapy of B-cell neoplasms. Clin Cancer Res. 2007 Sep 15;13(18 Pt 2):5556s-5563s. doi: 10.1158/1078-0432.CCR-07-1167. PMID 17875789